CLINICAL TRIAL: NCT04990778
Title: An Open Label, Phase II Investigator-Initiated Study of Venetoclax and Eprenetapopt (APR-246) in Previously Treated Relapsed/Refractory Patients With Mantle Cell Lymphoma (MCL)
Brief Title: Venetoclax and Eprenetapopt for the Treatment of Relapsed of Refractory Mantle Cell Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1325; NCI-2021-05596 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1325 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Recurrent Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — eprenetapopt; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (eprenetapopt, venetoclax) (Experimental): Patients receive eprenetapopt IV over 6 hours on days 1-4 and venetoclax PO QD. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Eprenetapopt; Drug: Venetoclax

INTERVENTIONS:
Drug: Eprenetapopt — Given IV
  Other Names: APR-246; PRIMA-1MET
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial investigates the effect of venetoclax and eprenetapopt in treating patients with mantle cell lymphoma that has come back (relapsed) or dose not respond to treatment (refractory). Chemotherapy drugs, such as venetoclax and eprenetapopt, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy (overall response rate) of the eprenetapopt plus venetoclax combination in relapsed refractory mantle cell lymphoma (MCL) patients (with/without TP53 aberrations).

SECONDARY OBJECTIVES:

I. To determine the safety profile of the eprenetapopt plus venetoclax combination in relapsed refractory MCL patients.

II. To evaluate the overall survival and progression-free survival of the eprenetapopt plus venetoclax combination in relapsed refractory MCL patients.

OUTLINE:

Patients receive eprenetapopt intravenously (IV) over 6 hours on days 1-4 and venetoclax orally (PO) once daily (QD). Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 months for 2 years, every 6 months for 5 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of mantle cell lymphoma in tissue biopsy and chromosome translocation t(11;14), (q13;q32) and/or overexpress cyclin D1 in tissue biopsy, cyclin D1 negative MCL (confirmed by hematopathology's are allowed and blastoid/pleomorphic morphology, complex karyotype are allowed)
* Patients must have relapsed or refractory MCL (irrespective of prior BTK inhibitor or anti CD19 chimeric antigen receptor T cell [CART] exposure)
* Prior exposure to venetoclax is allowed as long as the patients had clear evidence of disease progression on venetoclax (alone or in combination with other therapy) and the maximum dose of venetoclax was =< 400 mg. Doses > 400 mg and progression on venetoclax are excluded
* Patients with known TP53 status (positive or negative) - confirmed by a pre-treatment biopsy a pre-treatment biopsy to be sent for TP53 sequencing and TP53 testing by fluorescence in situ hybridization (FISH) and TP53 by immunohistochemistry (IHC) from hem-path to the hem-pathology and get the TP53 status before starting the study as a part of screening. To send bone marrow (BM) for TP53 assessment if it is involved by MCL > 10% instead
* TP53 mutation positive by IHC (>= 50%) in MCL cells and/or TP53 deletion by FISH in bone marrow (BM) or in tissues and/or del17p in karyotype or TP53 deletion positive by FISH in BM/involved tissue with MCL or presence of somatic TP53 mutations by next generation sequencing (NGS) or whole exome sequencing (WES) and TP53 wild type or mutation-negative status are allowed
* High risk MCL (blastoid/pleomorphic histology, high Ki-67 [>= 50%], TP53/NOTCH1/2, NSD2, CYCLIN D1, BIRC3 mutated, complex karyotype, Bulky disease > 5 cm, FISH positive for TP53 or MYC from involved tissues, high risk Mantle Cell Lymphoma International Prognostic Index [MIPI] score)
* Understand and voluntarily sign an Institutional Review Board (IRB)-approved informed consent form
* Age from >= 18 years at the time of signing the informed consent
* Patients must have bi-dimensional measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
* Absolute neutrophil count (ANC) > 1,000/mm^3

  * If bone marrow and spleen are involved, the counts of ANC will not be limited
* Platelet count >= 100,000/mm^3

  * If bone marrow and spleen are involved, the counts of platelets will not be limited
* Prothrombin time (or international normalized ratio) and partial thromboplastin time not to exceed 1.2 times the institution normal range (patients with an elevated prothrombin time and known lupus anticoagulant may be eligible for participation after consulting the medical monitor)
* Platelet count >= 100, 000/mm^3
* Absolute neutrophil count (ANC) >= 1000/mm^3 unless cytopenia is clearly due to marrow involvement from MCL
* Total hemoglobin >= 9 g/dL (without transfusion support within 2 weeks of screening);

  * If any of the above-mentioned cytopenias (a-c) are present due to significant BM involvement (requiring transfusion or granulocyte colony-stimulating factor [G-CSF] support) MCL patients may proceed with enrollment after discussion with the PI or designee. Cytopenias may not be due to evidence of myelodysplastic syndrome (MDS) or hypoplastic BM
* Creatinine clearance >= 30 mL/min (by Cockcroft-Gault method)
* Total serum bilirubin =< 1.5 x upper limit of normal (ULN) unless due to Gilbert's syndrome, non-Hodgkin lymphoma (NHL) organ involvement, controlled immune hemolysis or considered an effect of regular blood transfusions
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 x ULN, unless due to NHL organ involvement
* Projected life expectancy of > 12 weeks
* Female patients must be surgically sterile, postmenopausal (for at least 1 year), or have confirmed negative results for a pregnancy test at screening, on a blood or urine sample obtained within 7 days prior to initiation of study treatment
* Women of childbearing potential and men with female partners of childbearing potential must be willing to use an effective form of contraception
* Patient enrolled into the eprenetapopt + venetoclax study should use an effective form of contraception for up to 30 days after the last dose of eprenetapopt in combination with venetoclax, whichever time period is longer. Recommended methods of highly effective birth control are:

  * Hormonal contraception (birth control pills, patches, or rings)
  * Intrauterine device (IUD)
  * Birth control injections
  * Double barrier methods (diaphragm with spermicidal gel or condoms with birth control foam)
  * Sterilization of participant or partner ("tubes tied" or vasectomy)
* Disease free of prior malignancies with exception of currently treated basal cell, squamous cell carcinoma of the skin, carcinoma "in situ" of the cervix or breast, or other malignancies in remission (including prostate cancer patients in remission from radiation therapy, surgery or brachytherapy), not actively being treated, with a life expectancy > 3 years. Principal investigator (PI) could use judgment in the best interests of patients

Exclusion Criteria:

* Known central nervous system (CNS) involvement by lymphoma. Patients with previous treatment for CNS involvement who are neurologically stable and without evidence of disease (as shown by magnetic resonance imaging [MRI] brain and/or cerebrospinal fluid [CSF] or clinical exam by neurologists may be eligible if a compelling clinical rationale is provided to Aprea pharma which is the supporting company and the institution is the investigational new drug [IND] sponsor)
* Any serious uncontrolled medical condition including but not limited to, uncontrolled hypertension, diabetes mellitus, active/symptomatic coronary artery disease, chronic obstructive pulmonary disease (COPD), renal failure, active infection, active hemorrhage, laboratory abnormality, or psychiatric illness that places the patient at unacceptable risk and would prevent the subject from signing the informed consent form
* Pregnant or lactating females
* Known human immunodeficiency virus (HIV) infection
* Patients with active hepatitis B infection (not including patients with prior hepatitis B vaccination; or positive serum Hepatitis B antibody. Active hepatitis B/C. Patients with prior exposure to hepatitis B (i.e. positive anti-hepatitis B CORE antibody) must demonstrate hepatitis B polymerase chain reaction (PCR) to be negative during screening period and undergo prophylaxis and monitoring for hepatitis B according to institutional guidelines. Known hepatitis C infection is allowed as long as there is no active disease and is cleared by gastrointestinal (GI) consultation
* Clinically significant cardiovascular diseases as determined after cardiology consultation, including uncontrolled or symptomatic arrhythmias, congestive heart failure or myocardial infarction within 6 months of screening or any class 3 (moderate) or 4 (severe) cardiac disease following the New York Heart Association classification, known left ventricular ejection fraction (LVEF) < 40%, history of familial long QT syndrome, Symptomatic atrial or ventricular arrhythmias not controlled by medications. Otherwise, significant screening electrocardiogram (ECG) abnormalities and/or pacemaker may be allowed after discussion with the PI and the cardiologist clearance
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction. Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal (GI) absorption of venetoclax
* With known allergies to xanthine oxidase inhibitors and/or rasburicase
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that, in the opinion of the investigator, may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study
* No concomitant anticancer therapies, immunotherapies, cellular, or radiotherapy. No major surgery within 3 weeks prior to first dose of study treatment. Washout period for chemotherapy is 14 days. Washout period for targeted agents is 2 weeks or 5 half-lives (t1/2) (whichever is shorter). Washout period for antibody-based immunotherapies or cellular therapies is 4 weeks. Washout period for radiotherapy is 7 days (limited field) and 28 days (extended field that includes BM). Washout period must be completed prior to any treatment administration
* Uncontrolled autoimmune hemolytic anemia (AIHA) or immune thrombocytopenia
* Consumption of grapefruit, grapefruit products, Seville oranges, or star fruit within 7 days of starting study treatment
* Concomitant steroids for disease related pain control are allowed at any dose but must be discontinued prior to any study treatment initiation. Chronic use of corticosteroids is allowed up to 20 mg prednisone daily for non-cancer related conditions at the time of study start
* History of allogeneic or autologous stem cell transplant (SCT) or CAR-T therapy within the last 30 days or with any of the following:

  * Active uncontrolled graft versus host disease (GVHD)
  * Cytopenias from incomplete blood cell count recovery post-transplant;
  * Need for anti-cytokine therapy for residual symptoms of neurotoxicity > grade 1 from CAR-T therapy
* Ongoing immunosuppressive therapy
* Known neurologic disorder or residual neurologic toxicities that may put patients at increased risk of neurologic toxicity in the opinion of the investigator
* Concomitant malignancies or previous malignancies with less than a 1-year disease-free interval at the time of signing consent. Subjects with adequately treated basal or squamous cell carcinoma of the skin, or adequately treated carcinoma in situ (e.g. cervix) may enroll irrespective of the time of diagnosis. Patients with controlled, advanced prostate cancer (not on active chemotherapy) are permitted
* Active uncontrolled systemic infection
* Received an investigational agent within 30 days or within 5 T1/2, whichever is shorter prior to the first dose of study treatment
* Current treatment with certain strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers and/or strong P-glycoprotein (P-gp) inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2023-03-24 (Estimated); Study Completion 2023-03-24 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (complete and partial responses) | At 16 weeks
  Will be based on Cheson, Lugano Classification 2014. Its associated exact 95% confidence interval will be presented.

SECONDARY OUTCOMES:
Complete response rate | through study completion, an average of 1 year
  Will be based on Cheson, Lugano Classification 2014. Its associated exact 95% confidence interval will be presented.
Progression free survival | through study completion, an average of 1 year
  Kaplan-Meier methodology will be utilized.
Duration of response (DOR) | From the date of achieving earliest response (complete response or partial response) to the date this response is not maintained
  Will be summarized by providing the median DOR together with associated 95% confidence interval, using Kaplan-Meier methodology.
Overall survival | From the date of treatment start to date of death or last follow up either on or off study
  Kaplan-Meier methodology will be utilized.
Frequency of adverse events | Up to study completion
  Will be assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Severity of adverse events | through study completion, an average of 1 year
  Will be assessed by NCI CTCAE version 5.0.
Relatedness of treatment-emergent adverse events | through study completion, an average of 1 year
  Will be assessed by NCI CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Luhua (Michael) Wang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States